CLINICAL TRIAL: NCT00226876
Title: Dreaming During Anaesthesia and Anaesthetic Depth
Status: Completed | Type: Observational
Sponsor: Melbourne Health (Other)
Collaborators: Australian and New Zealand College of Anaesthetists (Other)
Responsible Party: Sponsor
Other Study IDs: 2005/016
Record Dates: First submitted 2005-09-26; First posted 2005-09-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-09

CONDITIONS: Anaesthesia
Keywords: dreaming; anaesthesia; electroencephalography; bispectral index; awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients commonly report that they have been dreaming when they awaken from general anaesthesia. Our hypothesis is that patients who report dreaming are less deeply anaesthetised during anaesthesia than patients who do not report dreaming. Depth of anaesthesia will be determined using a processed electroencephalographic monitor (called the BIS monitor).

DETAILED DESCRIPTION:
In this study, we will record the depth of anaesthesia during surgery with the BIS monitor and then interview patients immediately upon emergence to determine whether they recall dreaming or not. The depth of anaesthesia of dreamers and non-dreamers will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* American Society of Anesthesiologists physical status 1-3
* Non-cardiac surgery under relaxant general anaesthesia
* Tracheal extubation planned at end of surgery

Exclusion Criteria:

* Inadequate English language skills (due to language barrier, cognitive deficit or intellectual disability)
* Major drug abuse or psychiatric condition
* Expected to be unable to co-operate or be available for followup

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients presenting for elective non-cardiac surgery
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2005-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Leslie, MD, Principal Investigator — Melbourne Health
Locations (3):
- Australia (3):
  - Royal Melbourne Hospital, Melbourne, Victoria
  - King Edward Memorial Hospital for Women, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia